CLINICAL TRIAL: NCT04837170
Title: Safety and Efficacy Evaluation of S（+）-Ketamine for Postoperative Acute Pain in Adults in Perioperative Settings: A Multicenter, Randomized, Open-label, Active Controlled Pragmatic Clinical Trial
Brief Title: Safety and Efficacy Evaluation of S (+) - Ketamine in Adults
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Jiangsu Provincial People's Hospital (Other); Beijing Hospital (Other Government); The Affiliated Hospital of Qingdao University (Other); Renmin Hospital of Wuhan University (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); Shengjing Hospital (Other); Southern Medical University, China (Other)
Responsible Party: Principal Investigator, Weidong Mi, Director of the Department of Anesthesiology, Chinese PLA General Hospital, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAFE-SK-A
Record Dates: First submitted 2021-04-06; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Postoperative Pain; Adults; Anesthesia
Keywords: S-ketamine,Esketamine,S (+) - ketamine; Acute Pain; Depression, Anxiety; Delirium; Hyperalgesia
MeSH Terms: conditions — Pain, Postoperative; Acute Pain; Depression; Anxiety Disorders; Delirium; Hyperalgesia | interventions — Ketamine; Esketamine

STUDY DESIGN:
Intervention Model Description: Experimental group : Control group=2:1
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- S (+)-Ketamine group (Experimental): Drug: Conventional therapy + S (+)-Ketamine In principle, there are no specific restrictions on the dosage, mode of administration, timing, and compatibility of S-ketamine hydrochloride injection,but the recommended dosage is given, which is lower than the dosage specified in the instructions.
  Recommended use and dosage of S (+)-Ketamine:
  1. Bolus intravenous injection before skin incision, the dose is 0.1~0.5 mg/kg;
  2. Bolus intravenous injection (dose 0.1~0.5 mg/kg) before skin incision +continuous intravenous infusion (dose of 0.1~0.25 mg/kg/h) during operation;
  3. Continuous intravenous infusion after surgery with a dose of 0.02~0.1 mg/kg/h for 24~48 h.
  Interventions: Drug: Conventional therapy + S (+)-Ketamine
- Control group (Active Comparator): Drug: Conventional therapy Receiving conventional therapy without S (+)-Ketamine hydrochloride injection. There is no restrictions in drugs, doses and incompatibility, the researchers can choose appropriate medication regimens based on clinical practice, but other NMDA receptor antagonists are not be allowed to use, such as dextromethorphan and amantadine.
  Interventions: Drug: Conventional therapy

INTERVENTIONS:
Drug: Conventional therapy + S (+)-Ketamine — Patients who undergo general anesthesia using S(+)-ketamine hydrochloride for anesthesia induction,maintenance or postoperative analgesia.
  Other Names: Conventional therapy + S-ketamine; Conventional therapy + Esketamine
  Arms: S (+)-Ketamine group
Drug: Conventional therapy — Receiving conventional therapy without S (+)-Ketamine hydrochloride injection. There is no restrictions in drugs, doses and incompatibility, the researchers can choose appropriate medication regimens based on clinical practice, but other NMDA receptor antagonists are not be allowed to use, such as dextromethorphan and amantadine.
  Other Names: Routine treatment
  Arms: Control group

SUMMARY:
A multicenter, randomized, open-label, active controlled pragmatic clinical trial that evaluates the safety and efficacy of S (+) -ketamine for postoperative acute pain in adults in perioperative settings.

DETAILED DESCRIPTION:
Patients often suffer acute pain after operation ，which may affect the recovery. Opioid such as morphine is the most commonly analgesic drugs, but opioid has many obviously adverse reactions ,for example respiratory depression,circulation inhibition,tolerance, addiction, nausea, vomiting, pruritus, etc. S (+) - ketamine has been described to decrease acute pain and opioid consumption,but it needs to confirm for chinese patients undergoing surgery.

Objective:Evaluate the efficacy and safety of S (+) - ketamine on acute perioperative pain for chinese adult patients,and look for the best dosage, mode of administration, timing, and compatibility ,as well explore the effect of S (+) - ketamine on postoperative delirium,anxiety ,depression and cognitive dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥18 years old;
* 2. Scheduled for elective digestive tract surgery, gynecological surgery, urological surgery, thoracic surgery, orthopedic limb surgery, orthopedic spine surgery or body surface surgery (thyroid surgery or breast surgery), head and neck surgery;
* 3. ASA score Ⅰ～Ⅲ;
* 4. The informed consent form was signed by the patients.

Exclusion Criteria:

* 1. The expected length of hospital stay of the patient is less than 48h;
* 2. Patients expected to be admitted to the ICU after surgery;
* 3. Patients expected to return to the ward with tracheal catheter after surgery;
* 4. Be allergic to S (+) - ketamine;
* 5. Patients with severe disorder of consciousness or mental system diseases (schizophrenia, mania, bipolar disorder, psychosis, etc.) or cognitive dysfunction;
* 6. Patients with a history of severe cardiovascular disease (congestive heart failure, severe angina attack, or unstable angina or myocardial infarction within 6 months);
* 7. Patients during pregnancy or lactation;
* 8. Patients with MMSE score <18 points;
* 9. Patients with any of the following contraindications of S (+) - ketamine:

  1. Patients with risk of serious rise of blood pressure or intracranial pressure;
  2. Patients with high intraocular pressure (glaucoma) or penetrating ocular trauma;
  3. Patients with poorly controlled or untreated hypertension (Resting systolic blood pressure greater than 180 mmHg, or resting diastolic blood pressure greater than 100mmHg);
  4. Patients with untreated or undertreated hyperthyroidism.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12000 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
The area under the broken line of NRS score | Hour 0-48 after surgery
  The score of Numerical Rating Scale(NRS) is 0-10, the higher the score, the more severe the pain.
Opioid consumption | Hour 0-48 after surgery
  Total opioid consumption(conversion to equivalent morphine)

SECONDARY OUTCOMES:
NRS pain scores | Hour 0-48 after surgery
  The score of Numerical Rating Scale(NRS) is 0-10, the higher the score, the more severe the pain.
Time of first rescue analgesia | Hour 0-48 after surgery
  The time from the end of the operation to the first rescue analgesics after the operation. Rescue analgesia refers to the analgesia according to the patient's requirements in addition to routine postoperative analgesia.
The incidence of rescue analgesia | Hour 0-48 after surgery
  The incidence of rescue analgesia within 48h after surgery
Recovery time | Day 0
  The time from the end of the operation to recovery(can be awakened)
The incidence of unexpected intraoperative events | Intraoperative
  Unexpected events during operation include intraoperative cough, laryngeal spasm, body movement, tachycardia,decreased oxygen saturation, respiratory depression, bradycardia, hypertension and hypotension.
The Patient Efficacy Questionnaire (IPOQ ) scores | Hour 48 after surgery
  Patient Efficacy Questionnaire (IPOQ ) scale include 13 questions , each question's score is 0-10 or 0-100%, it involves postoperative pain, mood and quality of life. The higher the score, the more severe the pain symptoms.
The incidence of adverse events after surgery | Hour 0-48 after surgery
  The incidence of adverse events from the end of the operation to 48h after surgery. Including nausea, vomiting, increased secretions, dizziness, oversedation, infection,anesthetic awareness, nightmares, restlessness, pruritus, disorientation, delirium, respiratory depression, diplopia, diarrhea, intestinal obstruction, urinary retention, gastroesophageal reflux, constipation, chills, hallucinations, etc.
Pharmacoeconomic indicators | Hour 48 after surgery
  Calculating incremental cost-effectiveness ratio （ICER）based on cost-effectiveness analysis.
Incidence of postoperative delirium | Hour 0-48 after surgery
  The Chinese version of the 3D-CAM scale is used for the diagnosis of delirium, and the assessment will be carried out at 24h, 48h and 72h after the operation. If the patient is discharged 72h after the patient is discharged, it may not be assessed.
Simple Mental State Examination (MMSE) Scale score | Hour 48 after surgery
  The total score of Simple Mental State Examination Scale (MMSE) is 30,the higher the score, the better the cognitive function.
Hospital Anxiety and Depression (HAD) Scale score | Hour 48 after surgery
  Hospital Anxiety and Depression Scale (HAD) includes anxiety measure(7questions,0-21pionts) and depression measure(7 questions,0-21pionts),the higher the score, the more severe thesymptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Weidong Mi, MD, Study Chair — Chinese PLA General Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang H, Duan CY, Huang WQ, Zhao P, Zhou LZ, Liu YH, Liu CM, Chu HC, Wang Q, Diao YG, Hua Z, Meng QT, Li H, Zhang XY, Mi WD, Chen PY. Perioperative intravenous S(+)-ketamine for acute postoperative pain in adults: study protocol for a multicentre, randomised, open-label, positive-controlled, pragmatic clinical trial (SAFE-SK-A trial). BMJ Open. 2021 Dec 16;11(12):e054681. doi: 10.1136/bmjopen-2021-054681. PMID 34916327